CLINICAL TRIAL: NCT00246233
Title: A Double-blind, Placebo-controlled, Randomized Trial to Evaluate the Safety, Tolerability and Efficacy of CONCERTA® (Methylphenidate Hydrochloride) Augmentation of SSRI/SNRI Monotherapy in Adult Patients With Major Depressive Disorder.
Brief Title: CONCERTA® (Methylphenidate Hydrochloride) as add-on Therapy in the Treatment of Adult Major Depressive Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006073
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Depressive Disorder, Major
Keywords: methylphenidate hydrochloride; oral tablets; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Methylphenidate

INTERVENTIONS:
Drug: methylphenidate

SUMMARY:
The purpose of this study is to evaluate the effects of the addition of CONCERTA® (methylphenidate hydrochloride, a central nervous system (CNS) stimulant) or placebo in adult outpatients with Major Depressive Disorder who are currently being treated with oral antidepressant medication (selective serotonin reuptake inhibitors or selective norepinephine reuptake inhibitors). The general symptoms of depression will be evaluated, as measured by the Montgomery Asberg Depression Rating Score (MADRS) on fatigue, energy, and overall severity of illness. The safety and tolerability of the CONCERTA® and antidepressant combination therapy will also be assessed.

DETAILED DESCRIPTION:
Patient response to antidepressant therapy is low and 10-30% of depressed patients fail to respond to antidepressant therapy and of those patients who do respond, 50-75% exhibit a partial response. Augmentation and combination therapy strategies have been used in depressed subjects to enhance antidepressant response in treatment-resistant patients, to achieve remission in partial responders and to accelerate response. Augmentation of an antidepressant with CONCERTA® is an area open to new exploration in the adult population. This is a randomised, double-blind, placebo-controlled, parallel group, multicentre trial. Qualified subjects will have a diagnosis of Major Depressive Disorder, currently treated with an antidepressant, and will have demonstrated an insufficient treatment response to at least one but not more than three antidepressants. Subjects will continue their current treatment with oral antidepressant medication (selective serotonin reuptake inhibitors or selective norepinephine reuptake inhibitors) and be randomised to either CONCERTA® 18 mg or placebo. During the titration phase, subjects will take one tablet for the first 5 days and then be titrated up to the next dose level every week (2 tablets, then 3 tablets). At Week 4 and Week 5, subjects should be at their optimal, stable dose of the study drug. The maximum dose level is CONCERTA® 54 mg or placebo (3 tablets). Following titration, there are 5 weeks of treatment. The primary efficacy outcome is the change in total Montgomery Asberg Depression Rating Scale (MADRS) score between the two groups from baseline to the final visit. MADRS is a clinician-rated scale consisting of 10 items designed to assess a range of depressive symptoms. Safety and tolerability of study drug will be based on adverse events and clinical laboratory tests, ECG, vital signs and physical examination. The study hypothesis is that when CONCERTA® is added to antidepressant therapy, there will be a rapid, tolerable and overall improvement in symptoms of depression, as measured by the total Montgomery Asberg Depression Rating Score (MADRS).

Subjects will be randomized to a once-daily starting dose of 18mg CONCERTA® or 1 tablet of placebo to be taken orally. Provided patients are tolerating the study medication, they will be titrated weekly. There are 3 weeks of titration and one dose reduction allowed. The maximum dose level is 54 mg per day (3 tablets). By week 4 and week 5, subjects should be at their optimal dose. Following titration, there are 5 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Currently having a Major Depressive Disorder episode without psychotic features
* Has had an inadequate response to at least one but not more than 3 antidepressants given for 4 weeks
* Is currently treated with an antidepressant for the past 4 weeks
* Has a Montgomery Asberg Depression Rating Scale (MADRS) total score greater than or equal to 20, lassitude score of greater than or equal to 2 and a suicidal thought score less than 4
* Has a Clinical Global Impression of Severity (CGI-S) score greater than or equal to 4

Exclusion Criteria:

* Has a current diagnosis of schizophrenia, bipolar disorder, dementia, psychosis, obsessive-compulsive disorder, post-traumatic stress disorder, panic disorder, Attention Deficit Hyperactivity Disorder (ADHD), anorexia nervosa and/or bulimia nervosa, or a history of ADHD, anorexia nervosa and/or bulimia nervosa
* Agitated during the current depressive episode
* Has significant abnormal personality traits, which could interfere with function
* Has a history of substance abuse and or dependence within 6 months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2005-06; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Change in total Montgomery Asberg Depression Rating Scale (MADRS) score between the two groups from baseline to the final visit.

SECONDARY OUTCOMES:
Safety and tolerability of study drug based on adverse events and clinical laboratory tests, ECG, vital signs and physical examination, finding changes from baseline to the final visit.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada

REFERENCES:
- [Result] Ravindran AV, Kennedy SH, O'Donovan MC, Fallu A, Camacho F, Binder CE. Osmotic-release oral system methylphenidate augmentation of antidepressant monotherapy in major depressive disorder: results of a double-blind, randomized, placebo-controlled trial. J Clin Psychiatry. 2008 Jan;69(1):87-94. doi: 10.4088/jcp.v69n0112. PMID 18312042
- See also: A double blind, randomized trial to evaluate the safety,tolerability and efficacy of CONCERTA® augmentation of SSRI/SNRI monotherapy in adult patients with Major Depressive Disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=368&filename=CR006073_CSR.pdf